CLINICAL TRIAL: NCT01855399
Title: Technologically Enhanced Coaching (TEC):A Program for Improving Diabetes Outcomes
Brief Title: Technologically Enhanced Coaching: A Program to Improve Diabetes Outcomes
Acronym: VA-TEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 12-412
Record Dates: First submitted 2013-05-13; First posted 2013-05-16 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-04

CONDITIONS: Diabetes
Keywords: Peer Support; Self Management; Health Disparities
MeSH Terms: conditions — Diabetes Mellitus | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer Coaching + Decision Aid (Experimental): All participants will be assigned to one of up to 87 peer coaches, who also are Detroit VA diabetes patients who previously had poor glycemic control but are currently in good control. After their baseline assessment, participants in both arms will receive information on their lab and blood pressure values and will be randomized to one of the two study arms. Participants in the TEC arm will be scheduled for an initial visit with their coach to review the decision aid, which has incorporated their personal baseline data.
  Interventions: Behavioral: Peer Coaching; Behavioral: Decision Aid
- Peer Coaching Alone (Active Comparator): Participants randomized to the 'print materials' group will be scheduled for an initial visit with their coach. The coach will then help them list questions and concerns they wish to discuss with their health care provider, practice raising their questions and concerns and develop an action plan to address barriers to self-management they have identified. During the next six months coaches in both arms will call their assigned peers once a week to provide support for their action steps.
  Interventions: Behavioral: Peer Coaching

INTERVENTIONS:
Behavioral: Peer Coaching — All participants will be assigned to a peer coach, who is a Detroit VA diabetes patient who previously had poor glycemic control but is currently in good control. Participants will receive information on their lab and blood pressure values and will be scheduled for an initial visit with their coach. The coach will then help them list questions and concerns they wish to discuss with their health care provider, practice raising their questions and concerns, and develop an action plan to address barriers to self-management they have identified. During the next six months, coaches will call their assigned peers once a week to provide support for their action steps.
Behavioral: Decision Aid — The iDecide tool is designed to present key tailored, evidence-based information on diabetes and diabetes treatments. Importantly for a peer support intervention, all content information will be provided through the tool, with the role of the peer mentor being to assist the participant to go through the program and participate in helping the patient formulate questions and concerns to discuss with their health care provider, to set their own behavioral goals and action steps, and to help the participant practice raising the issues they plan to discuss with their health care provider.
  Other Names: TEC
  Arms: Peer Coaching + Decision Aid

SUMMARY:
Peer support programs have been demonstrated to improve glycemic control among Veterans with poor control. This program will expand on this success by putting innovative tools in the hands of Veteran diabetes patients. Veteran coaches who have demonstrated effective control of their own diabetes will be trained to use communication skills to guide their peers through a diabetes education and decision aid. This tool, which is an iPad application, draws the patient in by showing them their personal risk and medication information derived from baseline labs and self-reported survey data. The tool encourages interaction by providing choices of materials to view, using audio-visual elements and incorporating a goal-setting process for developing self-management action steps and questions to discuss with their doctor at their next clinic visit. Ongoing weekly contact between the Veterans is supported by a confidential phone system.

DETAILED DESCRIPTION:
Peer mentoring and support models have been found in two recent VA Randomized Controlled Trials (RCTs) to be more effective than usual care, financial incentives, and usual nurse care management to improve glycemic control in high-risk Veteran patients with poor glycemic control. Such models are important complements to provision of care by formal health care providers as they provide sustained, flexible between-visit support. Peer supporters and coaches can be trained in effective behavioral approaches to support other Veterans' self-management behaviors. Such supporters, however, necessarily lack the content expertise to help Veterans make informed treatment decisions and set health goals with their health care providers. Accordingly, in a recent study the investigators developed and tested a tailored, interactive computer-based tool with diabetes and medication information embedded in the tool's software that peer coaches and other outreach workers can employ to facilitate discussions with patients. Such tailored, interactive tools have been found to be more effective than generic educational and decision support tools in improving clinical and patient-centered outcomes. Moreover, these tools could enhance the sustainability and effectiveness of coaching programs to better prepare patients to set self-management goals and action plans, and to discuss treatment options with their health care providers. With VA support and input from Veterans, the investigators adapted the tailored, interactive computer-based tool for use with and by Veterans with diabetes. The investigators now propose to incorporate this tool into a peer mentor-led diabetes self-management coaching program among predominantly African American Veterans with poor glycemic control at the Detroit VA, a VA health system with high rates of poor risk factor control among diabetes patients. The investigators propose to evaluate this Technology-Enhanced Coaching (TEC) program. Specifically, the investigators propose to:

Aim 1: Test the effectiveness of a technology-enhanced peer coaching (TEC) program in improving glucose control relative to peer coaching without technology enhancement; and, also test the effectiveness of peer support compared to observed usual care. For the "usual care" observed group, the investigators will use electronic health record data to measure A1c levels.

Aim 2: Assess the impact of the intervention on key patient-centered outcomes, including patients' satisfaction and involvement with care, perceived social support, diabetes-specific quality of life, and medication adherence.

Aim 3: Identify patient characteristics associated with engagement in the intervention and mediators and moderators of the intervention's impact on patient outcomes.

In summary, the TEC program builds on the demonstrated strengths of peer support models and of tailored, interactive decision support tools in improving diabetes self-management and outcomes. This study will test incorporation of tailored interactive educational tools into a peer coaching model found in prior VA RCTs to be effective in improving diabetes outcomes.

The tools tested in the proposed intervention will be disseminated for use in other VA sites through a tool kit with training and support materials. Because the intervention addresses barriers to disease management for chronically ill patients, physicians, and case managers, the study may have broader impact on management practices for other chronic illnesses.

ELIGIBILITY:
Inclusion Criteria:

* one hospitalization with a diabetes-related ICD-9 code
* two outpatient visits with a diabetes-related ICD-9 code
* at least one prescription for a glucose control medication (insulin or oral agents) or monitoring supplies.
* [70] Potential participants must also have their most recent A1c in the prior 6 months be at least 8.0% if age < 70 or at least 8.5% if age 70+).

Exclusion Criteria:

* Using ICD-9 diagnostic codes, the investigators will exclude patients if they have an active substance abuse disorder or serious psychiatric illness:

  * PTSD
  * bipolar disorder
  * dementia
  * schizophrenia
  * or personality disorders
* We will then send names of the patients to their primary care providers to identify any patients who they do not recommend inviting to participate in the program.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. E. Michele Heisler, MD MPA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turner CD, Lindsay R, Heisler M. Peer Coaching to Improve Diabetes Self-Management Among Low-Income Black Veteran Men: A Mixed Methods Assessment of Enrollment and Engagement. Ann Fam Med. 2021 Nov-Dec;19(6):532-539. doi: 10.1370/afm.2742. PMID 34750128

RESULTS

PARTICIPANT FLOW:
Groups:
- Coaching With Decision Aid-TEC: All participants will be assigned to one of up to 87 peer coaches, who also are Detroit VA diabetes patients who previously had poor glycemic control but are currently in good control. After their baseline assessment, participants in both arms will receive information on their lab and blood pressure values and will be randomized to one of the two study arms. Participants in the TEC arm will be scheduled for an initial visit with their coach to review the decision aid, which has incorporated their personal baseline data.
  The coach will then help them list questions and concerns they wish to discuss with their health care provider, practice raising their questions and concerns and develop an action plan to address barriers to self-management they have identified. During the next six months coaches will call their assigned peers once a week to provide support for their action steps.
- Coaching Without the Decision Aid- Print Materials: Participants randomized to the 'print materials' group will be scheduled for an initial visit with their coach to review usual print diabetes education materials.
  The coach will then help them list questions and concerns they wish to discuss with their health care provider, practice raising their questions and concerns and develop an action plan to address barriers to self-management they have identified. During the next six months coaches in both arms will call their assigned peers once a week to provide support for their action steps.
Period: 6 Month
Arm/Group | Coaching With Decision Aid-TEC | Coaching Without the Decision Aid- Print Materials
Started | 146 | 144
Completed | 126 | 129
Not Completed | 20 | 15
Not completed — Lost to Follow-up | 12 | 9
Not completed — Withdrawal by Subject | 8 | 6
Period: 12 Month
Arm/Group | Coaching With Decision Aid-TEC | Coaching Without the Decision Aid- Print Materials
Started | 126 | 129
Completed | 119 | 118
Not Completed | 7 | 11
Not completed — Lost to Follow-up | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coaching With Decision Aid-TEC | Coaching Without the Decision Aid- Print Materials | Total
Number analyzed (Participants) | 146 | 144 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.7) | 62.1 (10.5) | 63.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 141 | 142 | 283
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 139 | 142 | 281
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 92 | 89 | 181
  White | 52 | 53 | 105
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
percent glycosylated hemoglobin [Mean (Standard Deviation); unit: percent glycosylated hemoglobin] | 9.1 (1.7) | 9.1 (1.7) | 9.1 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Glycosylated Hemoglobin
Description: Percent glycosylated hemoglobin is measured at baseline, 6 months, and 12 months to test the effectiveness of a technology-enhanced peer coaching (TEC) program in improving glucose control relative to peer support alone.
Time Frame: 6 Month
Measure: Mean (Standard Deviation); unit: Percent glycosylated hemoglobin
Groups:
- Peer Coaching + Decision Aid: All participants will be assigned to a peer coaches, who also is a Detroit VA diabetes patients who previously had poor glycemic control but is currently in good control. After their baseline assessment, participants will receive information on their lab and blood pressure values and will be scheduled for an initial visit with their coach to review the decision aid, which has incorporated their personal baseline data. The coach will then help them list questions and concerns they wish to discuss with their health care provider, practice raising their questions and concerns and develop an action plan to address barriers to self-management they have identified. During the next six months, coaches will call their assigned peers once a week to provide support for their action steps.
- Peer Coaching Alone: Participants will be scheduled for an initial visit with their coach to review usual print diabetes education materials. The coach will then help them list questions and concerns they wish to discuss with their health care provider, practice raising their questions and concerns and develop an action plan to address barriers to self-management they have identified. During the next six months, coaches will call their assigned peers once a week to provide support for their action steps.
Arm/Group | Peer Coaching + Decision Aid | Peer Coaching Alone
Number analyzed (Participants) | 121 | 122
Percent glycosylated hemoglobin | 8.38 (1.7) | 8.39 (1.7)

ADVERSE EVENTS:
Time Frame: 3 Years: September 2014 to September 2017
Arm/Group | Coaching With Decision Aid-TEC | Coaching Without the Decision Aid- Print Materials
All-Cause Mortality (participants affected / at risk) | 0/146 | 0/144
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/144
Other Adverse Events (participants affected / at risk) | 0/146 | 0/144

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2012-06-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT01855399/Prot_000.pdf
  • Statistical Analysis Plan (2012-06-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT01855399/SAP_001.pdf